CLINICAL TRIAL: NCT03572634
Title: A Combined Phase 1/2 Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of TP-0903 in Patients With Previously Treated Chronic Lymphocytic Leukemia (CLL)
Brief Title: Phase 1/2 Study of TP-0903 (an Inhibitor of AXL Kinase) in Patients With Previously Treated CLL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Given the extensive time projected to conclude the study hypothesis, it is no longer feasible to include this study of TP-0903.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-0903-102
Record Dates: First submitted 2018-05-21; First posted 2018-06-28 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Chronic Lymphocytic Leukemia; CLL; SLL; Small Lymphocytic Lymphoma
Keywords: Tolero; Phase 1/2; First in human; Previously treated Chronic Lymphocytic Leukemia (CLL); Previously treated Small Lymphocytic Lymphoma (SLL); AXL inhibitor; Cancer; Advanced Cancer; Relapsed / Refractory CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Recurrence | interventions — dubermatinib

STUDY DESIGN:
Intervention Model Description: Adult patients with CLL/SLL who:
  are intolerant to, or have had progressive disease on B-cell receptor antagonists, BCL-2 antagonists or other investigational treatments for CLL/SLL (Group 1-TP 0903 monotherapy); or have progression of disease on ibrutinib, yet the treating provider considers continuation of ibrutinib therapy to be in the best interest of the patient (Group 2-TP-0903 and ibrutinib combination therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1-TP 0903 monotherapy (Experimental): Adult patients with CLL/SLL who:
  are intolerant to, or have had progressive disease on B-cell receptor antagonists, BCL-2 antagonists or other investigational treatments for CLL/SLL
  Interventions: Drug: TP-0903
- Group 2-TP-0903 and ibrutinib combination therapy (Experimental): Adult patients with CLL/SLL who:
  have progression of disease on ibrutinib, yet the treating provider considers continuation of ibrutinib therapy to be in the best interest of the patient
  Interventions: Combination Product: TP-0903 and ibrutinib combination therapy

INTERVENTIONS:
Drug: TP-0903 — Monotherapy: PHASE 1: TP-0903 will be a 25 mg flat dose. The study drug will be administered orally once daily for 28 days (each cycle is 28 days; no drug-free period).
  Patients may continue to receive TP-0903 in 28-day cycles at the same dose given during Cycle 1 until they experience unacceptable toxicity or unequivocal disease progression. No intrapatient escalation of the TP-0903 dose is permitted.
  PHASE 2: The starting dose of TP-0903 will be the RP2D determined during Phase 1. TP 0903 will be administered orally at a fixed dose once daily for 28 days (each cycle is 28 days; no drug-free period) with repeated cycles permitted until a patient experiences unacceptable toxicity or unequivocal disease progression.
  Arms: Group 1-TP 0903 monotherapy
Combination Product: TP-0903 and ibrutinib combination therapy — Combination therapy: PHASE 1: TP-0903 and ibrutinib combination therapy: The starting dose of TP-0903 will be a 20 mg flat dose. TP-0903 will be administered orally once daily for 28 days (each cycle is 28 days; no drug-free period). Patients will also receive ibrutinib at the same dose that they were receiving immediately prior to study enrollment.
  Patients should continue with the combination of ibrutinib and TP-0903 for at least 3 months after study start.
  PHASE 2: The starting dose of TP-0903 will be the RP2D determined during Phase 1. Patients will also receive ibrutinib at the same dose that they were receiving immediately prior to study enrollment. Both TP 0903 and ibrutinib will be administered orally at fixed doses once daily for 28 days (each cycle is 28 days; no drug-free period).
  Arms: Group 2-TP-0903 and ibrutinib combination therapy

SUMMARY:
TP-0903 is an inhibitor of AXL kinase. TP-0903 has shown potent inhibition of AXL kinase and other TAM family members in a biochemical kinase assay. TP-0903 demonstrates corresponding activity in cancer cell lines and mouse xenograft efficacy models. TP-0903 is shown to block cancer cell epithelial-to-mesenchymal transitions. AXL was identified as a potential therapeutic target in chronic lymphocytic leukemia (CLL). TP 0903 was shown to induce apoptosis in CLL B-cells taken directly from patients.TP-0903 was equally potent against CLL cells regardless of risk-factor.

TP-0903 is a novel oral inhibitor that targets AXL kinase and reverses the mesenchymal phenotype associated with advanced cancers. TP-0903 has demonstrated profound single agent activity in CLL B cells taken directly from patients even if the patient has high risk factors (ie, 17p/P53 deletions) or progressed on other agents (ie, ibrutinib). TP-0903 is currently being evaluated in patients with refractory solid tumors (TP-0903-101). This proposed study is designed to identify the maximum tolerated dose (MTD), safety profile and recommended Phase 2 dose (RP2D) of TP-0903 in patients with previously treated CLL. Treatment cycles may be repeated if the patient continues to show benefit and if TP-0903 is reasonably well tolerated.

The study will investigate the safety, pharmacokinetics, pharmacodynamics, and clinical activity of TP-0903.

DETAILED DESCRIPTION:
This is a combined Phase 1/2 study of oral TP-0903 in patients with previously treated CLL/SLL. In both Phase 1 and Phase 2, study participants will be assigned to one of two defined patient groups:

* Group 1 (TP-0903 monotherapy): Patients with CLL/SLL who are intolerant to, or have progressed on, B-cell receptor antagonists and/or BCL-2 antagonists
* Group 2 (TP-0903 and ibrutinib combination therapy): Patients with CLL/SLL who have progressed on ibrutinib yet the treating provider considers continuation of ibrutinib therapy to be in the best interest of the patient.

Both groups of patients will be treated identically with TP 0903 and will undergo the same study assessments.

Phase 1 Patients will be enrolled in Group 1 and Group 2 in cohorts of 3 to 6 patients simultaneously. Group 2 will start at one dose level below the Group 1 starting dose. In each group, escalation of the TP-0903 dose will follow a standard 3+3 design with sequential cohorts of three patients treated with incrementally higher doses of TP 0903 until a dose-limiting toxicity (DLT) is observed and the maximum tolerated dose (MTD) is established. In the absence of DLTs, the dose will be increased using a modified Fibonacci dose escalation scheme.

Once the MTD or preliminary RP2D is identified, an expansion cohort of up to 6 patients will be enrolled in each patient group to confirm safety/suitability of the preliminary RP2D, to collect additional biomarker data, and to further explore efficacy.

It is expected that up to 27 patients will be enrolled in each patient group for a total of up to 54 patients (TP-0903 monotherapy and combination therapy with ibrutinib).

Additional dose levels, schedules, or disease indications of TP 0903 may be explored, as appropriate, based on the modulation of key biomarkers and the safety profile and clinical signals of activity.

Phase 2 In Phase 2, patients will be enrolled in Group 1 (TP 0903 monotherapy) and Group 2 (TP-0903 combination therapy with ibrutinib) based on the Simon 2 stage design. In Stage 1, up to 13 patients will be enrolled into each patient group (total of 26 patients). If there are no responses among these 13 patients in each group, the study will be stopped. Otherwise, Stage 2 will open to enroll 14 additional patients in each group for a total of 27 patients per group. If 4 or more responses are observed among 27 patients, the conclusion will be that the study treatment is worthy of further investigation.

If both patient groups enroll through Stage 2, it is anticipated that the total enrollment for Phase 2 will be 54 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years old
2. Have an established, pathologically confirmed diagnoses of CLL/ Small Lymphocytic Lymphoma (SLL) requiring therapy according to the 2018 IWCLL guidelines
3. Have received at least one prior therapy for CLL/SLL and can be classified in one of two patient groups:

   * Group 1 (TP-0903 monotherapy): Patients with CLL/SLL who are intolerant to, or have progressed on B-cell receptor antagonists and/or BCL-2 antagonists or other investigational treatments for CLL/SLL
   * Group 2 (TP-0903 and ibrutinib combination therapy): Patients with CLL/SLL who have progressed on ibrutinib, yet the treating provider considers continuation of ibrutinib therapy to be in the best interest of the patient
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2
5. Have adequate hematologic function:

   * Absolute neutrophil count (ANC) ≥500/µL
   * Platelet count ≥30,000/µL
   * Hemoglobin ≥8 g/dL in the absence of transfusions within the previous 2 weeks
6. Have adequate organ function:

   * Creatinine clearance ≥30 mL/min
   * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) level ≤2.5 × upper limit of normal (ULN)
   * Have a total bilirubin level ≤1.5 × ULN (unless secondary to Gilbert syndrome, hemolysis, or leukemia)
7. Have acceptable coagulation status:

   • Activated partial thromboplastin (aPTT) and prothrombin time (PT) ≤1.5 × ULN
8. Have a negative pregnancy test (if female of childbearing potential)
9. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an effective method of contraception (hormonal or barrier method of birth control, or abstinence) prior to study entry and for the duration of study participation and for at least 30 days after the last study drug dose. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Have read and signed the Institutional Review Board (IRB) approved informed consent form (ICF) prior to any study related procedure. (In the event that the patient is rescreened for study participation or a protocol amendment alters the care of an ongoing patient, a new ICF must be signed.)
11. Are able to comply with the requirements of the entire study

Exclusion Criteria:

1. Have undergone prior autologous or allogeneic stem cell transplant within ≤3 months, have not recovered from transplant associated toxicities, or requires graft versus host immunosuppressive therapy
2. Have known central nervous system (CNS) involvement
3. Have Richter's transformation of CLL
4. Have received any monoclonal antibody therapy directed at treatment of the patient's malignancy within 2 weeks prior to anticipated first dose
5. Have received any anticancer therapy including chemotherapy, radiotherapy, or an investigational anticancer drug within less than 5 half lives of the last dose of that treatment

   • This exclusion criterion is not applicable to patients requiring continuation on ibrutinib. (Note: Certain patients with a rapidly rising white blood cell count while on ibrutinib may need to remain on this drug for medical reasons. These patients will need to be approved by the Medical Monitor and treated in accordance with the protocol.)
6. Have received >20 mg/day of prednisone and 0.1 mg/day of mineralocorticoids within 7 days prior to anticipated first dose
7. Have a corrected QT interval of >450 msec (males) and >470 msec (females) using Fridericia's correction formula
8. Have a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, or cardiovascular disease or any other medical condition that, in the opinion of the Investigator, would adversely affect his/her participation in the study
9. Are pregnant and/or nursing, or refuse to use appropriate contraceptives during the course of the study and for at least 30 days after the last dose of study drug
10. History of another malignancy in the last 5 years except for the following adequately treated:

    * Local basal cell or squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix or breast
    * Papillary, noninvasive bladder cancer
    * Early stage prostate cancer for which observation is clinically indicated
    * Other Stage 1 or 2 cancers currently in complete remission
    * Any other cancer that has been in complete remission for 2 years or surgically cured. Medical Monitor may be contacted for additional determination of acceptable prior cancer history
11. Have known gastrointestinal disorders (eg, malabsorption syndrome), complications (eg, dysphagia), or surgery that could make consumption or absorption of oral medications problematic
12. Have an uncontrolled systemic infection (viral, bacterial, or fungal) or fever and neutropenia within 7 days prior to anticipated first dose
13. Have active and uncontrolled autoimmune cytopenias for 2 or more weeks including autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura (ITP)
14. Have received prior therapy with an AXL inhibitor
15. Have exhibited allergic reactions to a similar structural compound, biological agent, or formulation
16. Are unwilling or unable to comply with procedures required in this protocol
17. Have a history of severe adverse reaction (eg. hypersensitivity reaction, anaphylaxis) to sulfonamides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Komarnitsky, Study Director — Sumitomo Pharma America, Inc.
Locations (6):
- United States (6):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University - St Louis, St Louis, Missouri
  - Cornell University, New York, New York
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients at 2 sites; 6 study sites were initiated; study sites were medical clinics
  Recruitment started: Jan 21, 2019 Recruitment ended: January 21, 2020
Pre-assignment Details: Group 1 (TP-0903 monotherapy): Patients with CLL/SLL who are intolerant to, or have progressed on, B-cell receptor antagonists and/or BCL-2 antagonists Group 2 (TP-0903 and ibrutinib combination). Group 2 will start at one dose level below the Group 1 starting dose.
Groups:
- TP-0903 Monotherapy (25mg Dose of TP-0903): Patients who are intolerant to, or have had progressive disease on B-cell receptor antagonists and/or BCL-2 antagonists or other investigational treatments. This represents phase I, phase II never occurred and dose escalation did not occur.
- TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903): Patients who have progression of disease on ibrutinib and the treating provider considers continuation of ibrutinib therapy to be in the best interest of the patient. This represents phase I, phase II never occurred and dose escalation did not occur.
Period: Overall Study
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903): Patients with CLL/SLL who had progressed on ibrutinib, yet the treating provider considers continuation of ibrutinib therapy to be in the best interest of the patient. This represents phase I, phase II never occurred and dose escalation did not occur.
- Total: Total of all reporting groups
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: PHASE 1: Incidence of Dose-limiting Toxicities (DLTs) and Treatment Emergent Adverse Events.
Description: A DLT is defined as a drug-related toxicity that is observed to occur within the first 28 days of treatment
Time Frame: 28 days
Population: Primary and secondary efficacy endpoints were not analyzed via statistical methods due to low enrollment in Phase 1 and no enrollment in Phase 2.
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: PHASE 2: ORR in the Two Defined Patient Groups According to Guidelines Set Forth by the 2018 IWCLL
Description: Objective Response Rate ([ORR], ie, rate of complete response [CR] plus rate of partial response [PR] in the defined patient groups according to guidelines set forth by the 2018 International Workshop on CLL (IWCLL)
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: PHASE 1: Area Under the Plasma Concentration-time Curve From Zero to Infinity of Oral TP-0903 in the Defined Patient Groups
Description: Blood samples will be collected from patients so that derived PK parameters by non-compartment analysis may be conducted on Cycle 1
Time Frame: 28 days
Population: The study was stopped prematurely due to low enrollment across the 6 investigative sites. Efficacy endpoints could not be reached, and PK and PD test results could not be evaluated due to low sample size.
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: PHASE 1: Peak Plasma Concentration (Cmax) of Oral TP-0903 in the Defined Patient Groups
Description: as for outcome 3
Time Frame: 28 days
Population: as for outcome 3
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: PHASE 2: To Determine the Duration of Response
Description: Time from tumor response to disease progression
Time Frame: 2 years
Population: The study was stopped prematurely due to early discontinuation of the study as a result of low enrollment. Efficacy endpoints could not be reached, and PK and PD test results could not be evaluated due to low sample size. 1 patient was enrolled in the Monotherapy group, 2 patients were enrolled in the Combination therapy group; 3 patients in total were enrolled in the study.
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: PHASE 2: Rate of Overall Survival
Description: The time from first dose to objective tumor progression or death
Time Frame: 2 years
Population: as for outcome 3
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were defined as all AEs that begin on or after the date of first dose of study drug. All patients in the study participated in Phase 1; a 30 day follow-up visit as part of the protocol noted patients undergo a safety evaluation in which the patient's condition during the 30 days after the last dose of study drug can be assessed. There is a visit window of up to 14 days after completion of 30 days from the last dose (ie, within 45 days after last dose).
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not related to the drug product.
Arm/Group | TP-0903 Monotherapy (25mg Dose of TP-0903) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TP-0903 Monotherapy (25mg Dose of TP-0903) (N=1) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903) (N=2)
Increased Alanine Aminotransferase and Aspartate Aminotransferase levels (Investigations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TP-0903 Monotherapy (25mg Dose of TP-0903) (N=1) | TP-0903 and Ibrutinib Combination Therapy (20 mg Dose of TP-0903) (N=2)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Geographic tongue with aphthous ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (3)
Pyrexia (General disorders) | 0 (0) | 1 (2)
Decreased bilirubin level (Investigations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased alkaline phosphatase level (Investigations) | 0 (0) | 1 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Lymphocyte Count Increase (Investigations) | 0 (0) | 1 (1)
Nail Infections (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased Alanine Aminotransferase (Investigations) | 0 (0) | 1 (1)
Increased Aspartate Aminotransferase (Investigations) | 0 (0) | 1 (1)
Dsypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (2)
Urinanry Incontience (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Worsening Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Worsening Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Worsening peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Worsening Intermittent constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped early (21 January 2020) due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03572634/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03572634/SAP_001.pdf